CLINICAL TRIAL: NCT01630122
Title: Molecular and Diagnostic Classification of Non-Small Cell Lung Cancer From Fine Needle Aspirates
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: IRB00020151; CCCWFU 97112 (Other: Wake Forest University Health Sciences)
Record Dates: First submitted 2012-06-15; First posted 2012-06-28 (Estimated); Last update posted 2018-07-03 (Actual); Status verified 2018-07

CONDITIONS: Non-Small Cell Lung Cancer
Keywords: Trans-thoracic Needle Biopsy (TNB); Endobronchial Ultrasound Guided Transbronchial Needle Aspiration (EBUS-TBNA); Trans-esophageal Ultrasound Scanning with FNA (EUS-FNA)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients newly diagnosed non small cell lung cancer: patients with presumed newly diagnosed non small cell lung cancer, where radiographic studies and clinical description favor a probable diagnosis of non small cell lung cancer

SUMMARY:
The goal of this study is to demonstrate the feasibility of using a novel, validated panel of Non-Small Cell Lung Cancer (NSCLC) histology-predictive genes (the "A/S signature) as a diagnostic tool for use with small-volume Fine Needle Aspirate (FNA) biopsies.

Objectives:

1. To establish FNA biopsy requirements for FNA-based subtype classification of NSCLC.
2. To define a "fixed statistical model" of histologic subtype prediction in NSCLC.

Study methods: To establish FNA biopsy requirements for gene expression-based subtype classification of NSCLC, patients with presumed newly diagnosed NSCLC, where radiographic studies and clinical description favor a probable diagnosis of NSCLC, will undergo FNA biopsy according to current standard techniques . For this part of the study, approximately 40 biopsies of confirmed NSCLC will be collected for analysis.

To define a fixed statistical model of histologic subtype prediction in NSCLC, we will prospectively collect 50 FNAs. These FNAs will represent Adenocarcinoma (AC) and Squamous Cell Carcinoma (SCC) cases at a ratio of approximately 1:1. Additional cases of not otherwise specified (NOS), should they be encountered, may also be collected for later analysis. FNA samples qualified based on cell number or ribonucleic acid (RNA) yield (depending on the findings of our primary objective)will be assayed on the QGS platform.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a diagnostic FNA by the following diagnostic modalities utilizing FNA: Trans-thoracic Needle Biopsy (TNB), Endobronchial Ultrasound Guided Transbronchial Needle Aspiration (EBUS-TBNA), Trans-esophageal Ultrasound Scanning with FNA (EUS-FNA).
* Patients must have radiographic evidence for presumed lung cancer or have a previously diagnosed NSCLC with potential recurrence. Patient undergoing FNA of potential NSCLC metastatic lesions are also included (e.g., patients with hepatic metastases).
* Age >18 years. Used to define adult age who can independently provide consent.
* Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

* Patients whose FNA biopsy is unable to provide subtype classification by pathology or is non-diagnostic.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Non-Probability Sample
Enrollment: 103 (Actual)
Dates: Start 2012-06 (Actual); Primary Completion 2015-08-18 (Actual); Study Completion 2015-08-18 (Actual)

PRIMARY OUTCOMES:
Use of Ribonucleic acid-based molecular signature of tumor samples obtained by fine needle aspirate to discriminate subtypes of tumors relevant to treatment and outcomes. | Day 1
  To test a an 8-gene panel's accuracy in discriminating Non-Small Cell Lung Cancer tumors subtypes that are relevant to treatment and expected outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: Jimmy Ruiz, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States